CLINICAL TRIAL: NCT01657955
Title: Study of Bendamustine Hydrochloride Injection in Previously Untreated Chronic Lymphocytic Leukemia Patients
Brief Title: Bendamustine Hydrochloride Injection for Previously Untreated Chronic Lymphocytic Leukemia
Acronym: CLL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Lanjin Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGN0117
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Lymphocytic Leukemia; Leukemia; Neoplasms
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Neoplasms | interventions — Bendamustine Hydrochloride; Chlorambucil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bendamustine Hydrochloride Injection (Experimental): d1-d2,i.v.gtt, 100mg/m2/d, 28 days per cycle, at most 6 cycles.
  Interventions: Drug: Bendamustine Hydrochloride Injection
- Chlorambucil (Active Comparator): d1-d2, d15-d16, p.o., 0.4mg/kg/day, 28 days per cycle, at most 6 cycles(if WBC≥4×109 /L at d12-d14 ); d1-d2, p.o., 0.4mg/kg/day, 28 days per cycle, at most 6 cycles(if WBC<4×109 /L at d12-d14 );
  Interventions: Drug: Chlorambucil

INTERVENTIONS:
Drug: Bendamustine Hydrochloride Injection
  Arms: Bendamustine Hydrochloride Injection
Drug: Chlorambucil
  Other Names: Leukeran
  Arms: Chlorambucil

SUMMARY:
The purpose of this study is to determine whether bendamustine is effective in the treatment of initial treatment of Chronic Lymphocytic Leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of CLL;
* No prior or no standard treatment for CLL;
* Binet stage B, C or symptomatic stage A;
* Needs treatment to control diseases;
* (Eastern Cooperative Oncology Group)ECOG performance status ≤ 2
* Life expectancy ≥3 months
* Written informed consent

Exclusion Criteria:

* Patients were diagnosed with or treated for malignant tumors other than CLL (including active central nervous system lymphoma) within one year prior to entering the study
* Transformation to Richter's syndrome, or prolymphocytic leukemia(PLL)
* Autoimmune hemolytic anemia requiring glucocorticoid therapy
* Autoimmune thrombocytopenia requiring glucocorticoid therapy
* Alanine aminotransferase(ALT)>3 times upper limits of normal value, Aspartate aminotransferase(AST)>3 times upper limits of normal value, Total bilirubin(TBIL)>2 times upper limits of normal value, serum creatinine>1.5 times upper limits of normal value;
* Other serious Concomitant diseases which affect participation of this study(uncontrolled diabetes, gastric ulcer, cardiac and pulmonary diseases, at active phases of autoimmune diseases;
* Serious or uncontrolled infections;
* Central nervous system dysfunction with clinical symptoms;
* Patients received major surgery within 30 days prior to study entry;
* Pregnant or lactating women
* Allergic to study drug or mannitol
* Participation in any other clinical trials within 3 months prior to study entry

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 24 months

SECONDARY OUTCOMES:
Progress free survival(PFS) | 24 months
Duration of Response (DR) | 24 months
Overall Survival(OS) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lu G Qiu, M.D., Principal Investigator — Hematologic Hospital of Chinese Academy of Medical Sciences
Locations (1):
- Hematologic hospital of Chinese academy of medical sciences, Tianjin, China

REFERENCES:
- See also: Related Info — http://lanjin.cn